CLINICAL TRIAL: NCT00172575
Title: Differentiation of Malig. & Ben. Solitary Pulm. Nodules & Prediction of Clin. Outcome Using Perfus. Analysis of DCEMRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701184
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2004-12

CONDITIONS: Lung Neoplasms
Keywords: Lung neoplasms; Magnetic resonance imaging
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of our study is to determine whether contrast-enhanced dynamic MRI (DCE MRI) analysis of tumor angiogenesis and perfusion can be used as a reliable modality to differentiate benign from malignant solitary pulmonary nodules (SPN) before surgical intervention, using kinetic model derived from DCE MRI, and further correlate if there is any positive correlation between angiogenesis factor (vascular endothelial growth factor VEGF, microvessel density MVD); and if the perfusion parameters from DCE MRI can predict patients' outcomes and survival.

DETAILED DESCRIPTION:
The solitary pulmonary nodule (SPN) is a common finding in chest radiography. Pulmonary nodules larger than 1cm indicative of malignancy or with indeterminate finding according to morphology criteria have to be defined by invasive methods such as biopsy or surgical excision, and benign pathology makes up 20-50% of those resected pulmonary lesions. The lesions not receiving surgical intervention often need imaging follow-up on a regular basis for a long period of time to monitor the stability of the finding.

There are many reports regarding the MRI perfusion analysis of neoplasms from many organs, including bone marrow, liver, breast, cervix, and they stressed not only on comparison between benignity and malignancy, but also on monitoring the treatment outcomes after neoadjuvant chemotherapy, radiation therapy or anti-angiogenic agent therapy [7-15]. Dynamic contrast-enhanced MRI (DCE MRI) is not a standard examination for SPN, but there have been some data regarding the differentiation between malignant and benign SPN using DCE MRI, with MRI offering higher specificity compared to dynamic CT scan [6, 7, 16]. It was also reported that DCE MRI could delineate kinetic and morphologic differences in tumor angiogenesis and perfusion characteristics between malignant and benign pulmonary lesions with relatively high accuracy [7, 16]. The purpose of our study is to determine whether DCE MRI analysis of tumor angiogenesis and perfusion can be used as a reliable modality to differentiate benign from malignant SPN before surgical intervention, using kinetic model derived from DCE MRI, and further correlate if there is any positive correlation between angiogenesis factor (vascular endothelial growth factor VEGF, microvessel density MVD); and if the perfusion parameters from DCE MRI can predict patients' outcomes and survival.

ELIGIBILITY:
Inclusion Criteria:

* patients who have solitary pulmonary nodules in CT

Exclusion Criteria:

* patients who don't fit the above inclusion criteria

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-12; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Pan-Chyr Yang, PhD, Study Director — National Taiwan University Hospital; Tiffany Ting-Fang Shih, MD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Schaefer JF, Vollmar J, Schick F, Vonthein R, Seemann MD, Aebert H, Dierkesmann R, Friedel G, Claussen CD. Solitary pulmonary nodules: dynamic contrast-enhanced MR imaging--perfusion differences in malignant and benign lesions. Radiology. 2004 Aug;232(2):544-53. doi: 10.1148/radiol.2322030515. Epub 2004 Jun 23. PMID 15215548
- [Background] Yi CA, Lee KS, Kim EA, Han J, Kim H, Kwon OJ, Jeong YJ, Kim S. Solitary pulmonary nodules: dynamic enhanced multi-detector row CT study and comparison with vascular endothelial growth factor and microvessel density. Radiology. 2004 Oct;233(1):191-9. doi: 10.1148/radiol.2331031535. Epub 2004 Aug 10. PMID 15304661